CLINICAL TRIAL: NCT00096681
Title: Protocol for Cross-Sectional Survey of Acid-Fast Bacilli (AFB) Smear Positive and/or Culture Positive Tuberculosis in the Masiphumelele Township
Brief Title: Prevalence of HIV and Tuberculosis in Masiphumelele Township, Cape Town, South Africa
Status: Completed | Type: Observational
Sponsor: CIPRA SA (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: James McIntyre, CIPRA SA
Other Study IDs: CIPRA-SA Project 3A; U19AI053217 (NIH); CIPRA; Project 3A
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Results first posted 2011-02-17 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to estimate the amount of HIV and tuberculosis (TB) infection in individuals 15 years and older in the Masiphumelele township of Cape Town, South Africa. Data collected in this study will be used to predict the effect of introducing anti-HIV therapy in this community.

DETAILED DESCRIPTION:
TB is the most common opportunistic infection among HIV infected people, and is the most common cause of death in HIV infected people in Africa. The Masiphumelele township of Cape Town, South Africa, with its high rates of TB and HIV, is representative of many poor communities of Africa. Via random sampling, this study will assess the prevalence of HIV and TB infections in the Masiphumelele township. Knowledge gained from this study will be used to predict if introducing antiretroviral therapy will reduce the prevalence of TB in this community.

Selection and enrollment of participants will last about 4 months. Potential participants will be visited in their homes by fieldworkers, who will explain the study. Participants will be invited to either go to the clinic on the day of the fieldworker's visit or to go on a different day. Participants who go to the clinic on the day of the visit will have two sputum samples collected with a nebulizer. Participants who do not go to the clinic on the visit day will be given a sputum sample bottle and will be asked to collect a sputum sample in the early morning the day before their clinic appointment. At the clinic appointment, another sputum sample will be collected from these participants. Direct smear acid-fast bacilli and Mycobacterium tuberculosis cultures will be done on both sputum samples. Participants who test positive for TB will be referred for TB treatment at the clinic. Participants will also be asked to complete a study questionnaire and will undergo an anonymous oral HIV test at the clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Masiphumelele township for at least 1 week prior to study entry
* Willing to provide informed consent
* Willing to comply with study requirements

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents of the Masiphumelele township of Cape Town, South Africa
Sampling Method: Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2005-02; Primary Completion 2005-08 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Gail Bekker, MBChB, FCP, PhD, Study Chair — Department of Medicine, University of Cape Town; James McIntyre, MBChB, MRCOG, Principal Investigator — University of the Witwatersrand and Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital

REFERENCES:
- [Background] Aaron L, Saadoun D, Calatroni I, Launay O, Memain N, Vincent V, Marchal G, Dupont B, Bouchaud O, Valeyre D, Lortholary O. Tuberculosis in HIV-infected patients: a comprehensive review. Clin Microbiol Infect. 2004 May;10(5):388-98. doi: 10.1111/j.1469-0691.2004.00758.x. PMID 15113314
- [Background] Badri M, Wilson D, Wood R. Effect of highly active antiretroviral therapy on incidence of tuberculosis in South Africa: a cohort study. Lancet. 2002 Jun 15;359(9323):2059-64. doi: 10.1016/S0140-6736(02)08904-3. PMID 12086758

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants From the Community: The number of participants from the community who attended the clinic for a once off study visit
Period: Overall Study
Arm/Group | Participants From the Community
Started | 762
Completed | 762
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants From the Community
Number analyzed (Participants) | 762
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 726
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 422
  Male | 340
Region of Enrollment [Number; unit: participants]
  South Africa | 762

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Microbiologically Confirmed Pulmonary Tuberculosis
Description: Confirmed Pulmonary Tuberculosis based on the sputum smear and culture results. The sputum sample was obtained at the once off study visit.
Time Frame: Pulmonary Tuberculosis diagnosed from sputum sample obtained at the study visit
Measure: Number; unit: Participants
Arm/Group | Participants From the Community
Number analyzed (Participants) | 762
Participants | 23

2. Secondary Outcome: Number of Participants With a Positive HIV Test
Description: Prevalence of HIV in the community based on a positive oral mucosal transudate sample obtained at the once off study visit.
Time Frame: HIV status at the time of the study visit
Measure: Number; unit: Participants
Arm/Group | Participants From the Community
Number analyzed (Participants) | 762
Participants | 174

ADVERSE EVENTS:
Arm/Group | Participants From the Community
Serious Adverse Events (participants affected / at risk) | 0/762
Other Adverse Events (participants affected / at risk) | 0/762

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes